CLINICAL TRIAL: NCT03958279
Title: Normal and Pathological Values of Postvoiding Residual Volume in Early Postpartum Period and Their Predisposing Factors (PAREZ - Partus - Residual Urine)
Brief Title: Normal and Pathological Values of Postvoiding Residual Volume in Early Postpartum Period and Their Predisposing Factors
Acronym: PAREZ
Status: Terminated | Type: Observational
Why Stopped: Due to covid pandemia related restrictions
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Other Study IDs: EC/002/2018/UNBRuzinov
Record Dates: First submitted 2018-11-06; First posted 2019-05-22 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Urinary Retention
Keywords: postvoiding residual volume; early postpartum period
MeSH Terms: conditions — Urinary Retention | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primipara giving birth: The investigators involve every primipara giving birth in a period of two years.
  Exclusion criteria:
  * a) Unwilling to participate
  * b) Minors (under 18 years old)
  * c) Foetus mortus or perinatal death of the newborn
  * d) Admission of the newborn to the ICU
  * e) Unfamiliar with slovak language
  * f) Multiple pregnancy
  Interventions: Diagnostic Test: Ultrasound measurement of residual volume in the urinary bladder; Diagnostic Test: Questionnaire

INTERVENTIONS:
Diagnostic Test: Ultrasound measurement of residual volume in the urinary bladder — Aim of this study is to asses post voiding residual volume by ultrasound scan 3th day after delivery with consecutive scan after 6 weeks, and determination of data dispersion among the population of primiparas.
Diagnostic Test: Questionnaire — Simple questionaire concerning voiding problems, infectious complications, medicaments and breastfeeding during puerperium period (6weeks)

SUMMARY:
Aim of this study is to asses post voiding residual volume by ultrasound scan 3th day after delivery with consecutive scan after 6 weeks, and determination of data dispersion among the population of primiparas. In women with excessive retention (+2SD), risk factors such as duration of labour, use of epidural analgesia, instrumental delivery, maternal birth injury and weight of the newborn will be noted down.

DETAILED DESCRIPTION:
Pregnancy itself and vaginal delivery are well known risk factors for pelvic floor dysfunction. The rise in progesterone related to pregnancy has an inhibitory effect on bladder smooth muscle - decreased smooth muscle tonus in lower urinary tract. Weight and pressure of pregnant uterus and loosening of some of the pelvic ligaments changes the statics of pelvic floor. In addition, delivery itself influence lower urinary tract; an overdistension of urinary bladder can occur easily, also as oedema of urethra or urethral hinge apparatus injury during "crowning" of the fetal head.

All of these factors can affect consecutive function of lower urinary tract right after delivery. It is known that in 1,5% of women giving birth, symptomatic urinary retention develop in early postpartum period, with necessity of insertion of an indwelling catheter. Discussed risk factors are: epidural analgesia, instrumental delivery and primiparity. The investigators can assume that every woman in early postpartum period has (to some extend) even in normal circumstances postvoiding residual volume. There is few evidence in a literature about this postpartum residual volume and its predisposing factors.

Postvoiding residual volume can be risk factor for postpartum urinary infection, which forms second largest part in infectious morbidity of women. By determination of risk factors (for increased post voiding residual volume) the investigators could narrow the group of women which necessitate increased attention in postpartal monitoring.

ELIGIBILITY:
Inclusion Criteria:

* The investigators involve every primipara giving birth at 2nd Department of Obstetrics and Gynecology, University Hospital Bratislava and Comenius University, Bratislava, Slovak Republic in a period of two years

Exclusion Criteria:

* Unwilling to participate
* Minors (under 18 years old)
* Foetus mortus or perinatal death of the newborn
* Admission of the newborn to the ICU
* Unfamiliar with slovak language
* Multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — primipara giving birth
Study Population: primipara giving birth
Sampling Method: Probability Sample
Enrollment: 930 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in postvoiding residual volume | 6 weeks
  Volume of remaining urine in the urinary bladder after micturition - assessed by ultrasound, third day after delivery, and 6 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Záhumenský, MD, PhD., Study Chair — Comenius University, Faculty of Medicine, 2nd Department of Obstetrics and Gynecology
Locations (1):
- 2nd Department of Obstetrics and Gynecology, University Hospital Bratislava and Comenius University, Bratislava, Slovak Republic, Bratislava, Slovensko, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided